CLINICAL TRIAL: NCT01806168
Title: The Role of Fast or Slow Repetitive Transcranial Magnetic Stimulation as Adjunct Therapy in Civilian Post-Traumatic Stress Disorder
Brief Title: rTMS in the Treatment of PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Peter Y Chan, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H12-01578; V12-01578 (Other: Vancouver Coastal Health Research Institute)
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: Post-traumatic stress disorder; Repetitive transcranial magnetic stimulation; Civilians; Neurostimulation; Dorsolateral prefrontal cortex
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-frequency (1 Hz) rTMS (Active Comparator): Low-frequency active stimulation over the right dorsolateral prefrontal cortex (DLPFC) on 5 consecutive days every week for 2 weeks, for a total of 10 therapy sessions, with 37.5 minutes per session.
  Interventions: Device: rTMS
- High-frequency (10 Hz) rTMS (Active Comparator): High-frequency active stimulation over the right dorsolateral prefrontal cortex (DLPFC) on 5 consecutive days every week for 2 weeks, for a total of 10 therapy sessions, with 37.5 minutes per session.
  Interventions: Device: rTMS
- Sham rTMS (Placebo Comparator): Sham stimulation over the right dorsolateral prefrontal cortex (DLPFC) on 5 consecutive days every week for 2 weeks, for a total of 10 therapy sessions, with 37.5 minutes per session.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Magstim Super Rapid-2
  Other Names: repetitive transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to assess the effects of repetitive transcranial magnetic stimulation (rTMS) in civilian patients with a confirmed diagnosis of post-traumatic stress disorder (PTSD). This research study will determine whether low-frequency (1 Hertz [Hz]) or high-frequency (10 Hz) rTMS over the right dorsolateral prefrontal cortex (DLPFC) has an effect on symptoms of PTSD compared to sham rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of PTSD as determined by a structured interview using the Mini International Neuropsychiatric Interview (MINI)
* no change in psychotropic medications within 4 weeks before the start of rTMS
* age > 19 years and < 70 years
* competency to give informed consent

Exclusion Criteria:

* any non-fixed metal object or implant (including cochlear implants) in brain, skull, scalp, or neck within 30 cm of the magnetic rTMS coil
* implantable devices, including cardiac pacemakers and defibrillators
* other contraindications to rTMS, including history of seizures (except childhood febrile seizures) or recent and unexplained syncope, first-degree relative with a history of epilepsy, treatment with a medication known to substantially decrease the seizure threshold, or pregnancy
* psychiatric diagnoses of psychosis or psychotic disorder (including psychotic depression), bipolar type I disorder, or organic mental disorders
* substance abuse/dependence within the past 3 months
* active suicidal risk as judged by the clinician
* borderline or antisocial personality disorder
* acute medical illness, including cancer
* any significant central nervous system disorder, such as brain mass, stroke, etc.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Ong, MD, FRCPC, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Rayani K, Grabovac A, Chan P, Montgomery S, Ghovanloo MR, Sacchet MD. Brain stimulation enhances dispositional mindfulness in PTSD: an exploratory sham-controlled rTMS trial. Front Psychiatry. 2025 Apr 29;16:1494567. doi: 10.3389/fpsyt.2025.1494567. eCollection 2025. PMID 40365001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the psychiatry outpatient and community programs of Vancouver Coastal Health between 2014 and 2018. Some participants were recruited after attending an outpatient psychoeducation group but had not received formal group therapy. All assessments and treatments took place at Vancouver General Hospital in Vancouver, British Columbia, Canada.
Pre-assignment Details: 46 patients were assessed for eligibility. 15 were excluded: 7 did not meet inclusion criteria and 8 declined to participate. The remaining 31 patients were enrolled and randomized to one of three conditions.
Period: Overall Study
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Started | 11 | 10 | 10
Received Allocated Intervention | 11 | 9 | 9
Completed | 10 | 9 | 7
Not Completed | 1 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS | Total
Number analyzed (Participants) | 11 | 9 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.5) | 43.5 (12.4) | 49.5 (6.9) | 43.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 7 | 24
  Male | 1 | 2 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11 | 9 | 9 | 29
Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) [Mean (Standard Deviation); unit: units on a scale] — The Clinician-Administered PTSD Scale-IV (CAPS-IV) is a semi-structured instrument that assesses the intensity, frequency, and severity of PTSD symptoms. It consists of 17 symptom items, each rated on a 0-4 scale for frequency and a 0-4 scale for intensity, with higher scores indicating greater frequency/intensity. The frequency and intensity scores are then summed to yield a total item severity score (range 0-8). The minimum score of the overall scale is 0 and maximum is 17*8=136, with higher scores indicating more severe symptoms.
  units on a scale | 72.27 (25.34) | 69.44 (18.29) | 55.22 (13.17) | 66.10 (21.35)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV)
Description: The Clinician-Administered PTSD Scale-IV (CAPS-IV) is a semi-structured instrument that assesses the intensity, frequency, and severity of PTSD symptoms. It consists of 17 symptom items, each rated on a 0-4 scale for frequency and a 0-4 scale for intensity, with higher scores indicating greater frequency/intensity. The frequency and intensity scores are then summed to yield a total item severity score (range 0-8). The minimum score of the overall scale is 0 and maximum is 17 items * maximum severity score of 8 = 136 (higher scores indicating more severe symptoms).
Time Frame: Endpoint (treatment end) (Week 2).
Population: Intention-to-treat population analysed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low-frequency (1 Hz) rTMS: Low-frequency active stimulation over the right DLPFC on 5 consecutive days every week for 2 weeks, for a total of 10 therapy sessions, with 37.5 minutes per session.
  rTMS: Magstim Super Rapid-2
- High-frequency (10 Hz) rTMS: High-frequency active stimulation over the right DLPFC on 5 consecutive days every week for 2 weeks, for a total of 10 therapy sessions, with 37.5 minutes per session.
  rTMS: Magstim Super Rapid-2
- Sham rTMS: Sham stimulation over the right DLPFC on 5 consecutive days every week for 2 weeks, for a total of 10 therapy sessions, with 37.5 minutes per session.
  rTMS: Magstim Super Rapid-2
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 9 | 9
units on a scale | 59.80 (35.83) | 74.00 (30.97) | 65.12 (14.97)
Statistical Analysis 1: Comparison: Low-frequency (1 Hz) rTMS vs High-frequency (10 Hz) rTMS vs Sham rTMS; Test type: Other; p = 0.046, Mixed Models Analysis
Statistical Analysis 2: Comparison: Low-frequency (1 Hz) rTMS vs Sham rTMS; Test type: Equivalence — a < 0.05; p = 0.021, t-test, 2 sided
Statistical Analysis 3: Comparison: High-frequency (10 Hz) rTMS vs Sham rTMS; Test type: Equivalence — a < 0.05; p = 0.65, t-test, 2 sided

2. Secondary Outcome: PTSD Checklist for Civilians (PCL-C)
Description: The PTSD Checklist for Civilians (PCL-C) is a standardised self-report rating scale for PTSD comprising 17 items that correspond to the DSM-V symptoms of PTSD. A total symptom severity score (range = 17-85) can be obtained by summing the scores from each of the 17 items that have response options ranging from 1 "Not at all" to 5 "Extremely".
Time Frame: Endpoint (Week 2).
Population: Intention-to-treat population analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 9 | 9
score on a scale | 48.10 (23.54) | 53.44 (22.80) | 52.14 (10.05)
Statistical Analysis 1: Comparison: Low-frequency (1 Hz) rTMS vs High-frequency (10 Hz) rTMS vs Sham rTMS; To test primary and secondary outcomes, we utilized intention to treat data and linear mixed models with a group random effect. Significance was set to a < 0.05; Test type: Other; p = 0.93, Mixed Models Analysis

3. Secondary Outcome: Hamilton Depression Rating Scale, 21-item Version (HDRS-21)
Description: A clinician-rated assessment of depression symptoms consisting of 21 items rated on a scale from 0 to 4, 0 to 2, or 0 to 3, with higher scores indicating greater symptom severity in all cases. Minimum score = 0; maximum score = 53 (scores > 23 are considered to be severe).
Time Frame: Endpoint (Week 2)
Population: Intent-to-treat population analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 9 | 9
score on a scale | 12.30 (8.42) | 11.22 (7.99) | 14.44 (3.32)
Statistical Analysis 1: Comparison: Low-frequency (1 Hz) rTMS vs High-frequency (10 Hz) rTMS vs Sham rTMS; Test type: Other; p = 0.18, Mixed Models Analysis

4. Secondary Outcome: Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR)
Description: A self-report scale to assess symptoms of depression consisting of 16 items, 9 of which contribute to a summed total score (i.e., only the highest score of items 1-4, 6-9, and 15-16 are counted). Scores range from 0-3, with higher scores indicating more severe symptoms. Total scores range from 0-27, with scores >= 21 considered very severe, 20-16 severe, 11-15 moderate, and 6-10 mild depression.
Time Frame: Endpoint (Week 2)
Population: Intent-to-treat population analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 9 | 9
score on a scale | 12.66 (6.63) | 15.00 (7.15) | 9.42 (4.68)
Statistical Analysis 1: Comparison: Low-frequency (1 Hz) rTMS vs High-frequency (10 Hz) rTMS vs Sham rTMS; Test type: Other; p = 0.54, Mixed Models Analysis

5. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: A self-report scale to assess symptoms of anxiety, consisting of 21 items scored on a scale from 0-3, with higher scores indicating more severe symptoms. Total scores range from 0-63, with scores >= indicating potentially concerning levels of anxiety.
Time Frame: Endpoint (Week 2)
Population: Intent-to-treat population analysed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 9 | 9
score on a scale | 24.70 (18.19) | 22.77 (18.78) | 28.14 (10.97)
Statistical Analysis 1: Comparison: Low-frequency (1 Hz) rTMS vs High-frequency (10 Hz) rTMS vs Sham rTMS; Test type: Other; p = 0.86, Mixed Models Analysis

6. Secondary Outcome: Generalized Anxiety Disorder (GAD-7) Scale
Description: A brief self-report scale to assess symptoms of anxiety, consisting of 7 items each scored on a scale from 0-3, with higher scores indicating more severe symptoms. Total scores range from 0-21, with scores 0-4 suggesting minimal anxiety, 5-9 mild, 10-14 moderate, and 15-21 severe anxiety.
Time Frame: Endpoint (Week 2)
Population: Intent-to-treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 9 | 9
score on a scale | 11.90 (7.03) | 8.50 (8.53) | 11.75 (5.62)
Statistical Analysis 1: Comparison: Low-frequency (1 Hz) rTMS vs High-frequency (10 Hz) rTMS vs Sham rTMS; Test type: Other; p = 0.4, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Low-frequency (1 Hz) rTMS | High-frequency (10 Hz) rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/11 | 0/9 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-frequency (1 Hz) rTMS (N=11) | High-frequency (10 Hz) rTMS (N=9) | Sham rTMS (N=9)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Several limitations to this study should be highlighted. The sample size was limited and retention within the sham treated group further limited statistical power, which increases the possibility of both type 1 and type 2 error.

We did not verify the integrity of blinding, and we did not use imaging to define treatment targets. These are methodological considerations that should be included in future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-12-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT01806168/Prot_SAP_ICF_000.pdf